CLINICAL TRIAL: NCT06921343
Title: Iron Deficiency Without Anemia in Children With Newly Diagnosed Celiac Disease: A Randomized, Open-Label, Controlled Trial.
Brief Title: Iron Deficiency in Pediatric Celiac Disease: Diet vs. Iron Supplementation Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaplan Medical Center (Other)
Collaborators: Schneider Children's Hospital (Other); Rambam Hospital, Haifa, Israel (Unknown); Meir Medical Center (Other); Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Tal Ben-Ami, Head of Pedatric Hematology Unit, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMC-25-0038
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Celiac Disease in Children; Iron Deficiency
Keywords: Celiac disease; Pediatric celiac disease; Iron deficiency; Ferritin levels; Gluten-free diet; Iron supplementation
MeSH Terms: conditions — Iron Deficiencies; Celiac Disease | interventions — Iron; Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Gluten-free diet + Oral Iron Supplementation Iron (III) Hydroxide Polymaltose (50 mg/5 mL) at a single dose of 6 mg/kg/day, maximum 100 mg/day, for 3 months
  Interventions: Drug: Iron (III) Hydroxide Polymaltose (50 mg/5 mL); Other: Gluten-free diet
- Control group (Active Comparator): Gluten-free diet
  Interventions: Other: Gluten-free diet

INTERVENTIONS:
Drug: Iron (III) Hydroxide Polymaltose (50 mg/5 mL) — Participants randomized to the intervention group will receive oral iron supplementation in addition to a gluten-free diet. The specific iron formulation used in this study is Iron (III) Hydroxide Polymaltose (50 mg/5 mL) at a dosage of 6 mg/kg/day, up to a maximum of 100 mg/day, for 3 months.
  The iron supplement will be given once daily, preferably on an empty stomach or with vitamin C-containing foods to enhance absorption. Parents/caregivers will be instructed on proper administration, and adherence will be monitored through weekly self-reported intake logs and pharmacy dispensing records.
  This intervention is specifically targeted at children with newly diagnosed celiac disease and iron deficiency without anemia.
  The study follows a non-inferiority design, comparing the effect of iron supplementation versus a gluten-free diet alone on ferritin levels.
  Arms: Intervention group
Other: Gluten-free diet — Participants in the control group will follow a strict gluten-free diet, the standard-of-care treatment for celiac disease. No iron supplementation will be given. Compliance will be monitored through self-reported adherence and TTG antibody levels at follow-up.

SUMMARY:
This study aims to understand how to best manage iron deficiency in children newly diagnosed with celiac disease. Many children with celiac disease have low iron levels, even if they do not have anemia. While some doctors recommend iron supplements, others believe that simply following a gluten-free diet may be enough to restore iron levels naturally.

In this study, children with newly diagnosed celiac disease and low iron levels (but normal hemoglobin) will be randomly assigned to one of two groups:

Gluten-Free Diet Only - No additional iron supplements Gluten-Free Diet + Iron Supplementation Researchers will compare iron store levels over one year to see if iron supplements provide any additional benefit beyond the gluten-free diet alone. The study will also track possible side effects of iron supplements, such as stomach discomfort.

This study will help doctors determine the best approach to managing iron deficiency in children with celiac disease, ensuring they receive the safest and most effective treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label, non-inferiority trial designed to evaluate the necessity of iron supplementation in children newly diagnosed with celiac disease and iron deficiency without anemia. The study will compare two treatment strategies:

Gluten-Free Diet Alone Gluten-Free Diet + Iron Supplementation The primary objective is to determine whether a gluten-free diet alone is sufficient to restore ferritin levels or if iron supplementation provides a significant additional benefit.

Study Design & Methods Eligible participants will be randomly assigned to one of the two treatment groups.

Ferritin levels will be monitored at baseline, 4 months, and 12 months to assess improvements.

The study will also evaluate patient adherence to a gluten-free diet and iron supplementation, quality of life, as well as the incidence of gastrointestinal side effects related to iron supplement use.

This study is expected to provide evidence-based guidance for the management of iron deficiency in pediatric celiac disease, addressing a gap in current clinical recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 18 months to 18 years
* Newly diagnosed with celiac disease (based on ESPGHAN guidelines)
* Ferritin levels below 15 ng/dL
* Normal hemoglobin, MCV, and MCH levels for age and sex

Exclusion Criteria:

* IgA deficiency preventing TTG antibody monitoring
* Potential celiac disease (positive serology with normal intestinal histology)
* Underlying diseases that may cause anemia (e.g., Inflammatory bowel disease, eosinophilic gastrointestinal disease, certain gastritis types)
* Diseases affecting iron absorption (e.g., Cystic Fibrosis)
* Congenital anemia (e.g., Thalassemia, hereditary spherocytosis)
* Prior iron supplementation (>14 days oral iron within 2 months or IV iron within 6 months before diagnosis)

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in ferritin levels from baseline to 12 months | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  This study measures the change in serum ferritin levels in children with newly diagnosed celiac disease and iron deficiency (without anemia) over a 12-month period. Participants will have their ferritin levels assessed at:
  Baseline (At Diagnosis) 4 Months 12 Months The primary objective is to determine whether the gluten-free diet alone leads to a ferritin level increase that is non-inferior to the increase seen in children receiving oral iron supplementation in addition to a gluten-free diet.

SECONDARY OUTCOMES:
Change in Anti-TTG antibody levels | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Measures the change in anti-TTG IgA antibody levels, which indicates adherence to a gluten-free diet and mucosal healing in celiac disease.
Self-reported adherence to gluten-free diet | Weekly (for intervention group up to 12 weeks), monthly (via phone, control arm, up to 12 weeks)), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Intervention group: Weekly parent-reported logs for 3 months
  Control group: Monthly telephone questionnaires for 3 months Adherence will be scored based on self-report of unintentional or intentional gluten ingestion on a scale (0-4)
Adherence to iron supplementation (intervention group only) | Weekly up to 3 months after enrollment
  Measures compliance with iron supplementation in the experimental group.
  Assessment Methods:
  Parental reporting via weekly logs Pharmacy refill records
Percentage of participants with ferritin ≥15 ng/mL at 12 Months | 12 months (±1 month) after enrollment
  Determines the proportion of participants who achieve normal iron stores (Ferritin ≥15 ng/mL) at the 12-month follow-up.
  Helps assess the effectiveness of the interventions in restoring iron stores.
Change in weight | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Evaluates weight patterns in children with celiac disease by measuring:
  Weight (kg)
Gastrointestinal symptoms evaluation | Weekly (Intervention Group Only up to 12 weeks)), 4 Months (±1 month), 12 Months (±1 month) after enrollment
  Symptoms recorded in a standardized questionnaire using units on a scale (0-4)
Evaluation of hemoglobin levels for anemia | 4 months (±1 month), 12 months (±1 month) after enrollment
  Monitor hemoglobin levels in both study groups to identify participants who develop anemia, which would necessitate early withdrawal from the study and initiation of iron treatment.
  Hemoglobin blood tests will be conducted at 4 months and 12 months for all participants.
  If a participant develops hemoglobin levels below age-adjusted reference values, the study protocol requires discontinuation from the trial and initiation of iron therapy as per clinical guidelines.
  The frequency of anemia-related study withdrawals will be documented and analyzed.
Association of H. pylori at diagnosis with GI symptoms | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Evaluate whether children with H. pylori-positive gastric biopsies at the time of celiac disease diagnosis experience a higher frequency or severity of gastrointestinal (GI) symptoms during follow-up compared to H. pylori-negative participants.
  GI symptoms will be assessed using standardized questionnaires with units on a scale (0-4)
Change in height | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Evaluates height patterns in children with celiac disease by measuring:
  height (cm)
Change in BMI | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Evaluates BMI patterns in children with celiac disease. Weight and height will be combined to report BMI in kg/m^2
Association of H. pylori at diagnosis with Ferritin levels over time | At baseline (Day 0), 4 months (±1 month), and 12 months (±1 month) after enrollment
  Assess whether the presence of H. pylori in gastric biopsies at the time of celiac disease diagnosis is associated with the trajectory of ferritin (ng/ml) levels from baseline through 12 months, in both the iron supplementation and diet-only groups.
Change in anti-TTG IgA antibody levels as an indicator of adherence to gluten-free diet | At 4 months (±1 month) and 12 months (±1 month) after enrollment
  Anti-TTG IgA levels in U/mL

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Assuta Ashdod Medical Center, Ashdod, Israel
  - Rambam Medical Center, Haifa, Israel
  - Meir Medical Center, Kfar Saba, Israel
  - Schneider Children's Medical Center, Petah Tikva, Israel
  - Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No
The study collects sensitive data on pediatric participants. Due to privacy concerns and limitations in obtaining broad consent for future use of individual-level data, IPD will not be shared.

REFERENCES:
- [Background] Ben-Ami T, Trotskovsky A, Topf-Olivestone C, Kori M. Iron deficiency without anemia in children with newly diagnosed celiac disease: 1-year follow-up of ferritin levels, with and without iron supplementation. Eur J Pediatr. 2024 Nov;183(11):4705-4710. doi: 10.1007/s00431-024-05721-1. Epub 2024 Aug 27. PMID 39190044